CLINICAL TRIAL: NCT03203733
Title: Cryoprotection of Chemotherapy-induced Oral Mucositis After Autologous Stem Cell Transplantation, a Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BraincoolUppsalaU
Record Dates: First submitted 2017-06-09; First posted 2017-06-29 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Cryotherapy Effect
Keywords: Oral Mucositis , cooling, cryotherapy
MeSH Terms: conditions — Stomatitis | interventions — Cryotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Cooral™' (Experimental): oral cooling with use of cooling device
  Interventions: Device: Cooral™
- cryotherapy (Active Comparator): Cryoterapy consists of ice cubes or crossed ice and used as standard treatment for oral cooling.
  Interventions: Other: cryotherapy

INTERVENTIONS:
Device: Cooral™ — An intraoral cooling device which is as effective as ice but with better patient comfort. The cooling device has the advantage that the water temperature can be modified. It enables that the unacceptable low temperatures that occur with ice cooling can be avoided.
  Arms: 'Cooral™'
Other: cryotherapy — Oral cooling by ice chips or crushed ice or ice pop
  Arms: cryotherapy

SUMMARY:
This study evaluates, among study patients with lymphoma or myeloma undergoing autologous SCT, whether cooling oral mucosa with a cooling device compared with ice cubes/crushed ice or ice pop succeeds in reducing the degree of oral mucositis (OM) according to the Oral Mucositis Assessment Scale (OMAS) total,degree of OM according to World Health Organisation (WHO), tolerability of either cooling method. The study is also aiming to , patients subjective experience of OM, rating of general quality of life and oral pain, number of days with total parenteral nutrition (TPN), number of hospital days, total dose of opioids, and C reactive protein during time in care.

Finally, the study aims to evaluate weight loss, Leukocyte particle concentration, number of days until bone marrow response, S-albumin, and body temperature.

DETAILED DESCRIPTION:
The degree of OM is assessed at eight intraoral locations, in accordance with the Oral Mucositis Assessment Scale (OMAS) (graded 0-3 for ulceration and 0-2 for erythema). 0 corresponds to "normal" while 3 and 2 are "sore >3 cm2" and "severe erythema" respectively. The assessment generates both an average for OMAS ulceration (0-3) and OMAS erythema (0-2) and a total average OMAS (0-5), which is the mean of both ulceration and erythema.

Besides OMAS, ulceration and erythema are also assessed with the WHO scale (graded 0-4) where 0 is "no mucositis" and 4 is "ulceration, total parenteral nutrition".

Assessment with OMAS and WHO is done by a dentist, blinded to treatment group, three times a week, for example, Monday, Wednesday, Friday, until discharge or at most day +28.Assessment with the WHO is also performed by nurses who are not blinded to the treatment group, three times a week.

Furthermore, the patients, after cooling ends, assess the tolerability of the respective cooling method with the aid of a questionnaire developed for the study. The questionnaire is intended to give some idea of any discomfort or side effects the patients feel as a result of the cooling method.

The patients assess their perception of oral problems daily with the aid of specific questions in a diary developed for the study. The questions are intended to give a picture of the effect of OM on the patient's general status.

General quality of life is assessed twice during the study period, before the start of treatment and at discharge, with a validated quality of life instrument.

Oral pain is assessed with a visual analog scale (VAS) with the extremes graded on a 10-figure scale (0-10) where 0 is "no pain" and 10 is "unbearable pain".

Information about total parenteral nutrition (TPN), number of hospital days, total dose of opioids, weight loss, and body temperature will be retrieved from patient records. Laboratory results of blood tests will be retrieved from each department's register of test results.

The result of the assessments is documented on sheets for the purpose in a patient's individual kardex.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 16 and 99 years of age diagnosed with lymphoma or myeloma
* Able to communicate in Swedish
* Treated with bis-chloroethylnitrosourea, etoposide, cytarabine, and cyclophosphamide(BEAC) or bis-chloroethylnitrosourea, etoposide, cytarabine, and melphalan (BEAM) (lymphoma diagnosis), melphalan (myeloma diagnosis), before stem cell transplantation (SCT)

Exclusion Criteria:

* Patients who do not understand oral and written information in Swedish.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
OM according to OMAS total during 28 days or until discharge | 28 days or until discharge
  Assesment with OMAS is done by a dentist blinded to treatment group, three times a week during 28 days or until discharge. Assessment with the not blinded to the treatment group, three times a week during 28 days or until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Garming Legert, Dentist, PhD, Principal Investigator — Section for Orofacial diagnosis and surgery, Karolinska University Hospital; Mats Jontell, dentist, Study Director — Oral Medicine Clinic, Department of Odontology, University of Gothenburg; Torbjörn Karlsson, MD physician, Principal Investigator — Section for Hematology & Coagulation, Uppsala University Hospital; PA Broliden, MD, PhD,, Principal Investigator — Hematology Center, M54, Karolinska University Hospital; Franz Rommel, physician, Principal Investigator — Section for Hematology, Linköping University Hospital; Erik Ahlstrand, physician, Principal Investigator — Section for Hematology, Örebro University Hospital
Locations (5):
- Rikshospitalet in Oslo, Oslo, Norway
- Sweden (4):
  - Linköping University Hospital, Linköping
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson DE, Bensadoun RJ, Roila F; ESMO Guidelines Working Group. Management of oral and gastrointestinal mucositis: ESMO Clinical Practice Guidelines. Ann Oncol. 2011 Sep;22 Suppl 6(Suppl 6):vi78-84. doi: 10.1093/annonc/mdr391. No abstract available. PMID 21908510
- [Background] Lalla RV, Bowen J, Barasch A, Elting L, Epstein J, Keefe DM, McGuire DB, Migliorati C, Nicolatou-Galitis O, Peterson DE, Raber-Durlacher JE, Sonis ST, Elad S; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2014 May 15;120(10):1453-61. doi: 10.1002/cncr.28592. Epub 2014 Feb 25. PMID 24615748
- [Background] Elting LS, Keefe DM, Sonis ST, Garden AS, Spijkervet FK, Barasch A, Tishler RB, Canty TP, Kudrimoti MK, Vera-Llonch M; Burden of Illness Head and Neck Writing Committee. Patient-reported measurements of oral mucositis in head and neck cancer patients treated with radiotherapy with or without chemotherapy: demonstration of increased frequency, severity, resistance to palliation, and impact on quality of life. Cancer. 2008 Nov 15;113(10):2704-13. doi: 10.1002/cncr.23898. PMID 18973181
- [Background] Naidu MU, Ramana GV, Rani PU, Mohan IK, Suman A, Roy P. Chemotherapy-induced and/or radiation therapy-induced oral mucositis--complicating the treatment of cancer. Neoplasia. 2004 Sep-Oct;6(5):423-31. doi: 10.1593/neo.04169. PMID 15548350
- [Background] Legert KG, Remberger M, Ringden O, Heimdahl A, Dahllof G. Reduced intensity conditioning and oral care measures prevent oral mucositis and reduces days of hospitalization in allogeneic stem cell transplantation recipients. Support Care Cancer. 2014 Aug;22(8):2133-40. doi: 10.1007/s00520-014-2190-7. Epub 2014 Mar 20. PMID 24647488
- [Background] Rubenstein EB, Peterson DE, Schubert M, Keefe D, McGuire D, Epstein J, Elting LS, Fox PC, Cooksley C, Sonis ST; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Clinical practice guidelines for the prevention and treatment of cancer therapy-induced oral and gastrointestinal mucositis. Cancer. 2004 May 1;100(9 Suppl):2026-46. doi: 10.1002/cncr.20163. PMID 15108223
- [Derived] Ibrahim A, Mahmoud D, Mavandadipur H, Walladbegi J. Interrater reliability in the assessment of oral mucositis among patients receiving high-dose chemotherapy: a multicenter comparison between specialized dentists and registered nurses. BMC Cancer. 2025 Dec 17;25(1):1874. doi: 10.1186/s12885-025-14670-3. PMID 41408611
- [Derived] Walladbegi J, Henriksson R, Tavelin B, Svanberg A, Larfors G, Jadersten M, Schjesvold F, Mahdi A, Garming Legert K, Peterson DE, Jontell M. Efficacy of a novel device for cryoprevention of oral mucositis: a randomized, blinded, multicenter, parallel group, phase 3 trial. Bone Marrow Transplant. 2022 Feb;57(2):191-197. doi: 10.1038/s41409-021-01512-6. Epub 2021 Nov 3. PMID 34728786
- [Derived] Walladbegi J, Svanberg A, Gellerstedt M. Protocol for a randomised controlled trial to study cryoprevention of chemotherapy-induced oral mucositis after autologous stem cell transplantation. BMJ Open. 2018 Oct 24;8(10):e021993. doi: 10.1136/bmjopen-2018-021993. PMID 30361399